CLINICAL TRIAL: NCT05483192
Title: Evaluation the Impact of Oral Dichrostachys Glomerata Extract (Dyglomera™) in Overweight and Obese Adults for Reducing Body Fat and Modulating Blood Parameters a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Impact of Oral Dyglomera™ on Body Fat and Blood Lipids of Overweight and Obese Adults
Acronym: Dyglomera
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gateway Health Alliance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/11/049204
Record Dates: First submitted 2022-07-19; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Body Fat Disorder
Keywords: Body fat; Dyglomera; Blood lipids

STUDY DESIGN:
Intervention Model Description: 12-week randomized, double-blind, placebo-controlled trial with subjects administered 400 mg per day of Dyglomera
Who Masked: Participant, Care Provider
Masking Description: To maintain double-blinding, in addition to the contents mentioned in the production/packaging and labeling of the products used in the human study, the allocation details of unique codes (information on blinding) for each group will be managed in a sealed state by the principal investigator. Except in cases where it is unavoidably necessary to read the code due to the occurrence of a serious adverse drug reaction*, it will not be disclosed until the end of the human study. In this human study, no unblinding will occur during the study. The investigator will supply the investigational products that match the randomization code assigned to the selected subject, and maintain blinding by using an extra (by unique code) when the investigational product is defective or damaged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison between placebo and active treatment (Placebo Comparator): 120 subjects were planned. Screening data was reviewed to determine subject eligibility. Subjects who met all inclusion criteria and none of the exclusion criteria were enrolled into the study.
  The following investigational products were used:
  * Test product: Dichrostachys glomerata extract (Dyglomera™) at a dose of 400 mg
  * Control product: Placebo at a dose of 400 mg Subjects were assigned to the test group or placebo group in random order. Each subject was administered a single 400 mg dose of Dyglomera or placebo once daily, before lunch or dinner. Measurements were taken at baseline and at the beginning of each of the 5 study visits.
  Interventions: Dietary Supplement: Oral Dyglomera
- Comparison of baseline to final outcome (Active Comparator): The effect of Dyglomera on body fat and blood parameters were compared at baseline and at the end of the intervention period.
  Interventions: Dietary Supplement: Oral Dyglomera

INTERVENTIONS:
Dietary Supplement: Oral Dyglomera — Measurement of body weight, waist circumference, hip circumference, waist to hip ratio, body mass index, body fat.
  Blood draw and measurement of blood total Cholesterol, HDL-cholesterol, LDL-cholesterol), ALT, AST, Fasting Blood Glucose, CRP, adiponectin, and leptin.
  Other Names: Placebo

SUMMARY:
The extract of Dichrostachys glomerata (DyglomeraTM), has been reported to be effective in weight reduction in obese patients with metabolic syndrome. This plant has been shown to have many biological properties and has been reported to have no toxic or adverse side effects in animals. The purpose of this human study was to prove that the effect of reducing body fat percentage (%) after 12 weeks of intake was superior to that of the control group.

DETAILED DESCRIPTION:
This is a 12-weeks randomized double-blind placebo controlled trial. 120 number of subjects are planned. Each subject will be administered a single dose of the investigational product once daily, before lunch or dinner, consisting each time of 400 mg of the test product or placebo. Subjects will be assigned to the test group or placebo group in random order. Evaluations will be taken at baseline and at the beginning of each of the 5 study visits.

Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

The following investigational products will be used:

* Test product: Dichrostachys glomerata extract (Dyglomera™) at a dose of 400 mg
* Control product: Placebo at a dose of 400 mg In this human study, starting with Visit 2, the duration of participation in the human study will be 12 weeks (84 days) in total. The study period will be planned to be 8 months from the date of approval of the human study. The screening visit of the first subject will be conducted at the MAX SPECIALTY HOSPITAL, and the first subject will be enrolled thereafter. The last subject will complete the study within about 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 19 to 65 years old,
* Patients with a BMI ranging between 25 and 34.9 kg/m2,
* Patients available for the entire period of study .

Exclusion Criteria:

* Patients that has an age below 19 years old and greater than 65 years old,
* Patients not available for the study period,
* Specific exclusion criteria included: morbid obesity (BMI > 34.9 kg/m2); diabetes mellitus requiring daily insulin management; pregnancy/lactation; active infection; and systemic disease such as HIV/AIDS, active hepatitis or clinical signs of active malignancy within the past 5 years. Other exclusion criteria will include having taken any other medications or any natural health product within 1 month prior to the screening visit.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Effect of Dyglomera on body fat of overweight and obese people | 12 weeks
  DEXA and impedance measurement of body fat

SECONDARY OUTCOMES:
Effect of Dyglomera on blood cholesterol levels of overweight and obese people | 12 weeks
  Blood assay to measure blood total cholesterol
Effect of Dyglomera on blood triglyceride levels of overweight and obese people | 12 weeks
  Blood assay to measure blood total triglycerides
Effect of Dyglomera on HDL-cholesterol levels of overweight and obese people | 12 weeks
  Blood assay to measure HDL-cholesterol
Effect of Dyglomera on fasting blood glucose levels | 12 weeks
  Blood assay to measure fasting blood glucose
Effect of Dyglomera on CRP levels of overweight and obese people | 12 weeks
  Blood assay to measure CRP
Effect of Dyglomera on ALT levels of overweight and obese people | 12 weeks
  Blood assay to measure ALT
Effect of Dyglomera on AST levels of overweight and obese people | 12 weeks
  Blood assay to measure blood AST
Effect of Dyglomera on leptin levels of overweight and obese people | 12 weeks
  Blood assay to measure leptin
Effect of Dyglomera on adiponectin levels of overweight and obese people | 12 weeks
  Blood assay to measure blood adiponectin
Effect of Dyglomera on blood insulin levels of overweight and obese people | 12 weeks
  Blood assay to measure insulin

CONTACTS AND LOCATIONS:
Locations (1):
- Max Super Specialty Hospital, New Delhi, Patparganj, India

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in the management of overweight and obese people. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)
URL: http://www.gha.org